CLINICAL TRIAL: NCT04015336
Title: A Phase II Study of E7 TCR T Cell Induction Immunotherapy for Stage II and Stage III HPV-Associated Oropharyngeal Cancer
Brief Title: E7 TCR Cell Induction Immunotherapy for Stage II and Stage III HPV-Associated Oropharyngeal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Logistical challenges
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Scott Norberg, D.O., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 190122; 19-C-0122
Record Dates: First submitted 2019-07-06; First posted 2019-07-11 (Actual); Results first posted 2022-02-01 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Papillomavirus Infections; Oropharyngeal Neoplasms
Keywords: T Cell Receptor; Fludarabine; Cyclophosphamide; Immunotherapy; Aldesleukin
MeSH Terms: conditions — Papillomavirus Infections; Oropharyngeal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 1-3x10^10 E7 T-Cell Receptor (TCR) T cells (Experimental): Up to 3x10^10 E7 T-Cell Receptor (TCR) T cells (based on the number of cells that can be generated in the shortened manufacturing process) will be administered intravenously over 20 to 30 minutes on day 0.
  Interventions: Biological: E7 T-Cell Receptor (TCR)

INTERVENTIONS:
Biological: E7 T-Cell Receptor (TCR) — The dose of E7 T-Cell Receptor (TCR) T cells will be 3 x 10^10 TCR+ T cells (unless fewer cells are generated) administered once.

SUMMARY:
Background:

The therapy used in this study is called E7 T-cell receptor (TCR) T cell therapy. This therapy is a type of treatment in which a participant's T cells (a type of immune system cell) are changed in the laboratory to attack cancer cells. This treatment might help people with human papillomavirus (HPV)-associated oropharyngeal cancer. Oropharyngeal cancer is a type of head and neck cancer that happens in the oropharynx (the part of the throat at the back of the mouth, including the soft palate, the base of the tongue, and the tonsils). Certain types of the HPV virus can cause this kind of cancer. This study is looking at treatments for cancer caused by HPV-16.

Objective:

The purpose of this study is to determine if E7 TCR T cells can be given safely without delaying standard treatment for HPV-16 associated oropharyngeal cancer. Standard treatment may be surgery or radiation therapy with chemotherapy.

Eligibility: People ages 18 and older with Stage II or III HPV-16 associated oropharyngeal cancer

Design:

Participants will be screened with HLA typing (a blood test needed for eligibility) and HPV testing of the cancer tumor (to determine if the cancer is HPV-16 positive). A new biopsy may be needed if tumor from an outside location is not available for HPV testing. Eligible participants will come to the National Institutes of Health (NIH) campus to have a screening evaluation which will include physical exam, review of medical history and current medications, blood and heart tests, imaging (X-ray, computed tomography (CT) scan, magnetic resonance imaging (MRI) or positron emission tomography (PET) scan), and evaluation of participant's veins that are used for drawing blood.

If the participant is eligible for the study based on the screening evaluation, they will have a baseline evaluation prior to receiving the experimental treatment. The baseline evaluation may include additional laboratory or imaging tests.

Participants will have a large intravenous (IV) catheter inserted into a vein to undergo a procedure called leukapheresis. Leukapheresis is the removal of the blood by a machine to collect specific blood cells. The remaining blood is returned to the body. This procedure is needed to collect the cells that will be modified to target the cancer. These cells will be grown in the lab and given back to the participant through an IV. It takes 11-15 days to grow the cells.

While the cells are growing, the participant will be admitted to the hospital about one week before cell infusion. They will receive 2 types of chemotherapy through an IV catheter over 5 days. The main purpose of the chemotherapy is to make the cells more effective in fighting the cancer tumors. The cells will be given through an IV catheter 1-3 days after the last dose of chemotherapy. Within 24 hours after the cell infusion, participants will be given a cell growth factor called aldesleukin through an IV. Aldesleukin is thought to help the cells live longer in the participant s body. Participants will recover in the hospital until they are well enough to go home. This is usually about 7-12 days after the cell infusion or last dose of aldesleukin.

Participants will have follow-up visits starting every 2 weeks after the date of cell infusion. These will be visits to monitor the safety of the treatment and to evaluate the response of the cancer to the treatment. These visits will continue if the cancer is shrinking. The participant will go back to their local cancer doctor for further care if the cancer stops shrinking, goes away completely or gets bigger.

Participants will have blood drawn periodically to test if the cells have grown or changed. These blood tests will take place immediately before the cells are given, and then at 3, 6, 12 months for the first year and then annually. These tests can be drawn locally and sent to the NIH. Participants will be asked to return to the NIH annually for a physical examination for 5 years after they receive the cells. After that time, participants will be asked to fill-out a questionnaire for the next ten years, for a total follow-up period of 15 years.

DETAILED DESCRIPTION:
Background:

* Human papillomavirus (HPV)+ oropharyngeal cancer is an increasingly common type of cancer that frequently affects young patients.
* The treatment for locoregionally advanced cancer carries substantial life-long morbidity.
* Although the overall prognosis for HPV+ oropharyngeal cancer is favorable, about 20 percent of patients with stage II disease and 35 percent of patients with stage III disease will die within five years.
* Induction therapy is an area of active study in this type of cancer. The aims of induction therapy are to reduce the risk of disease recurrence and potentially to permit the study of de-intensified definitive treatment of locoregional disease.
* E7 T-cell receptor (TCR) T cells, administered as a single infusion, have demonstrated safety and clinical activity in treatment-refractory metastatic HPV+ cancers.

Objectives:

-To determine the feasibility of systemic treatment with E7 TCR T cells for stage II or stage III HPV+ oropharyngeal cancer.

Eligibility:

* Patients greater than or equal to 18 years old with stage II or stage III HPV+ oropharyngeal cancer.
* The cancer must be HPV16+ and patient must be human leukocyte antigen-A (HLA-A) 02:01+ HLA type.
* Patients must be treatment-naive.

Design:

* This is a phase II, single arm, feasibility study of induction E7 TCR T cell therapy.
* Patients will receive a conditioning regimen of cyclophosphamide and fludarabine, a single infusion of E7 TCR T cells, and systemic aldesleukin.
* Patients will be referred for standard of care definitive therapy (chemoradiation or surgery) at the time of maximum tumor response

ELIGIBILITY:
* INCLUSION CRITERIA:
* Histologically or cytologically confirmed stage II or stage III (American Joint Committee on Cancer (AJCC) 8th edition) oropharyngeal squamous cell carcinoma that has not been treated.
* Human papillomavirus 16 (HPV16)+ tumor and human leukocyte antigen A (HLA-A) 02:01+ HLA type (HLA-A 02 is also acceptable for determination of eligibility).
* Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria.
* Patient age 18 and older. Because no dosing or adverse event data are currently available on the use of E7 T-cell receptor (TCR) T Cells in patients <18 years of age, children are excluded from this study. This reflects the age range of patients with the disease being studied.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* Women of child-bearing potential must have a negative pregnancy test because E7 TCR T Cells have unknown potential for teratogenic or abortifacient effects. Women of child-bearing potential are defined as all women who are not post-menopausal or who have not had a hysterectomy. Postmenopausal will be defined as women over the age of 55 who have not had a menstrual period in at least 1 year.
* The effects of E7 TCR T Cells on the developing human fetus are unknown. For this reason and because the chemotherapy agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (intrauterine device, hormonal or barrier method of birth control; abstinence; tubal ligation or vasectomy) prior to study entry and for four months after treatment. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Seronegative for human immunodeficiency virus (HIV) antibody. The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune-competence and thus be less responsive to the experimental treatment.
* Seronegative for hepatitis B antigen and hepatitis C antibody. If hepatitis C antibody test is positive, then the patient must be tested for the presence of antigen by Reverse transcription polymerase chain reaction (RT-PCR) and be hepatitis C virus ribonucleic acid (HCV RNA) negative.
* Must be willing to participate in Gene Therapy Long Term Followup Protocol, which will follow patients for up to 15 years per Food and Drug Administration (FDA) requirements.
* Patients must have organ and marrow function as defined below:

  * leukocytes- greater than or equal to 3,000/mcL
  * absolute neutrophil count- greater than or equal to 1,500/mcL
  * platelets- greater than or equal to 100,000/mcL
  * hemoglobin- greater than or equal to 9.0 g/dL
  * total bilirubin- within normal institutional limits except in patients with Gilbert's Syndrome who must have a total bilirubin < 3.0 mg/dL
  * Aspartate aminotransferase (AST) Serum glutamic oxaloacetic transaminase(SGOT)/Alanine transaminase (ALT) Serum glutamic pyruvic transaminase(SGPT)-Serum ALT/AST < 2.5 times upper limit of normal (ULN)
  * creatinine clearance- Calculated creatinine clearance (CrCl) >50mL/min/1.73m(2) for patients with creatinine levels above institutional normal (by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation)
* Ability of subject to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* Patients who are receiving any other investigational agents.
* History of severe allergic reactions attributed to compounds of similar chemical or biologic composition to agents used in study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations at the time of treatment that would limit compliance with study requirements.
* There is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with E7 TCR T Cells. For this reason, women may not breastfeed while receiving study treatment and for one year after the study treatment ends. These potential risks may also apply to other agents used in this study.
* Patients with any form of systemic immunodeficiency, including acquired deficiency such as human immunodeficiency virus (HIV) or primary immunodeficiency such as Severe Combined Immunodeficiency Disease, are ineligible. The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the treatment.
* Current use of immunosuppressive medication, EXCEPT for the following:

  * Intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection);
  * Systemic corticosteroids at physiologic doses less than equal to 10 mg/day of prednisone or equivalent;
  * Steroids as premedication for hypersensitivity reactions (e.g., computed tomography (CT) scan premedication)
* Patients with autoimmune diseases such as Crohn's disease, ulcerative colitis, rheumatoid arthritis, autoimmune hepatitis, autoimmune pancreatitis, or systemic lupus erythematosus. Hypothyroidism, vitiligo and other minor autoimmune disorders are not exclusionary.
* Patients with a second active invasive cancer are not eligible if it may confound assessment of response to the current therapy.
* Patients who do not have a local physician to provide standard therapy post treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott M Norberg, D.O., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared as follows: Coded, linked data in an National Institutes of Health (NIH)-funded or approved public repository, coded, linked data in Biomedical Translational Research Information System (BTRIS), and identified or coded, linked data with approved outside collaborators under appropriate agreements.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Before publication and at the time of publication or shortly thereafter.
Access Criteria: Clinical Trials.gov, Biomedical Translational Research Information System (BTRIS), approved outside collaborators under appropriate individual agreements, and publication and/or public presentations.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2019-C-0122.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1-3x10^10 E7 T-Cell Receptor (TCR) T Cells
Started | 1
Completed | 0
Not Completed | 1
Not completed — Participant signed consent and was later deemed a screen failure. Participant was not treated | 1

BASELINE CHARACTERISTICS:
Arm/Group | Arm 1-3x10^10 E7 T-Cell Receptor (TCR) T Cells
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.1 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Fraction of Participants Who Can Receive Induction Therapy With E7 T-Cell Receptor (TCR) Cells Without Failing the Feasibility Criteria
Description: Fraction of participants who can receive induction therapy with E7 T-Cell receptor (TCR) cells without failing the feasibility criteria with 95% confidence intervals. The feasibility criteria is defined as follows, 1) delivery of the E7 TCR T Cell induction therapy without an increase in tumor T or N stage between baseline and the last response assessment before referral for definitive treatment, 2) initiation of definitive therapy without a delay in treatment related to toxicity of the induction therapy, and 3) if any participant starts the conditioning regimen chemotherapy but does not receive the E7 TCR T Cells it will be considered a feasibility failure. Failure by one criterion will be scored as a feasibility failure.
Time Frame: 3 months
Population: Data was not collected for this outcome measure. This outcome measure was not done because the single enrolled participant signed consent and was later deemed a screen failure, thus was unable to receive induction therapy with E7 TCR cells. Participant was not treated and the study was terminated due to logistical challenges.
Arm/Group | Arm 1-3x10^10 E7 T-Cell Receptor (TCR) T Cells
Number analyzed (Participants) | 0

2. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Description: Here is the number of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 9 days.
Population: This outcome measure was not done because the participant was not evaluable for toxicity since the toxicity evaluation begins at the time of induction therapy. The participant was never treated with induction therapy.
Arm/Group | Arm 1-3x10^10 E7 T-Cell Receptor (TCR) T Cells
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: The participant was not evaluable for toxicity since the toxicity evaluation begins at the time of induction therapy. The participant was never treated with induction therapy.
Arm/Group | Arm 1-3x10^10 E7 T-Cell Receptor (TCR) T Cells
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2020-11-04): https://cdn.clinicaltrials.gov/large-docs/36/NCT04015336/Prot_SAP_000.pdf
  • Informed Consent Form: Screening consent (2021-01-05): https://cdn.clinicaltrials.gov/large-docs/36/NCT04015336/ICF_001.pdf
  • Informed Consent Form: Treatment consent (2021-01-05): https://cdn.clinicaltrials.gov/large-docs/36/NCT04015336/ICF_002.pdf